CLINICAL TRIAL: NCT01272063
Title: Measurement and Analysis of Macular Retinal Pigment Epithelium (RPE) Elevations With Cirrus HD-OCT vs. Color Fundus Photography
Status: Completed | Type: Observational
Sponsor: Carl Zeiss Meditec, Inc. (Industry)
Collaborators: DataMed Devices Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HD-OCT-DR-2010-1
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Drusen Stage Macular Degeneration
Keywords: Drusen; Dry AMD; OCT; Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dry AMD with macular drusen: Patients diagnosed with dry AMD with macular drusen

SUMMARY:
The objective of this study is to compare the areas designated as elevated retinal pigment epithelium (RPE) by the Cirrus HD-OCT versus those designated as drusen on color fundus photographs (CFPs).

DETAILED DESCRIPTION:
This is a prospective, multiple site study. Ocular history and examination will be conducted on consented subjects to determine further participation in the study. Subjects qualified to continue will undergo color fundus photography and imaging of their study eye using the Cirrus HD-OCT.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 50 years of age or older diagnosed to have dry AMD with macular drusen.
* Drusen should not be combined with other lesions such as geographic atrophy (GA) or choroidal neovascularization.
* Able and willing to make the required study visits.
* Able and willing to give consent and follow study instructions.

Exclusion Criteria:

* History of retinal surgery, laser photocoagulation, and/or radiation therapy to the eye.
* Evidence of other retinal diseases of the eye, including wet AMD, diabetic retinopathy, diabetic macular edema, or significant vitreomacular traction upon dilated examination, or upon evaluation of retinal photos.
* Thick media opacity or inability to fixate that precludes obtaining acceptable scans.
* Concomitant use of hydrochloroquine and chloroquine.
* Unable to make the required study visits.
* Unable to give consent or follow study instructions.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To compare area measurements of elevated RPE as observed in the Cirrus HD-OCT versus those designated as drusen on color fundus photographs. | Study was released before December 1, 2012

SECONDARY OUTCOMES:
To describe the clinical factors that affected the automated segmentation of elevated RPE by the Cirrus HD-OCT. | Study was released before December 1, 2012

OTHER OUTCOMES:
To describe the qualitative similarities and differences between the areas designated as elevated RPE by the Cirrus HD-OCT versus those designated as drusen on color fundus photographs. | Study was released before December 1, 2012

CONTACTS AND LOCATIONS:
Overall Officials: Philip Rosenfeld, MD, Principal Investigator — Bascom Palmer Eye Institute; Carmelina Gordon, MD, Principal Investigator — TLC Eyecare and Laser Center; Eugene Lit, MD, Principal Investigator — East Bay Retina Consultants; Brandon Lujan, MD, Principal Investigator — West Coast Retina
Locations (4):
- United States (4):
  - East Bay Retina, Oakland, California
  - West Coast Retina, San Francisco, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - TLC Eyecare and Laser Centers, Lansing, Michigan

REFERENCES:
- [Background] Klein R, Cruickshanks KJ, Nash SD, Krantz EM, Nieto FJ, Huang GH, Pankow JS, Klein BE. The prevalence of age-related macular degeneration and associated risk factors. Arch Ophthalmol. 2010 Jun;128(6):750-8. doi: 10.1001/archophthalmol.2010.92. PMID 20547953
- [Background] Varma R, Foong AW, Lai MY, Choudhury F, Klein R, Azen SP; Los Angeles Latino Eye Study Group. Four-year incidence and progression of age-related macular degeneration: the Los Angeles Latino Eye Study. Am J Ophthalmol. 2010 May;149(5):741-51. doi: 10.1016/j.ajo.2010.01.009. PMID 20399926
- [Background] Yi K, Mujat M, Park BH, Sun W, Miller JW, Seddon JM, Young LH, de Boer JF, Chen TC. Spectral domain optical coherence tomography for quantitative evaluation of drusen and associated structural changes in non-neovascular age-related macular degeneration. Br J Ophthalmol. 2009 Feb;93(2):176-81. doi: 10.1136/bjo.2008.137356. Epub 2008 Aug 12. PMID 18697811
- [Background] Jain N, Farsiu S, Khanifar AA, Bearelly S, Smith RT, Izatt JA, Toth CA. Quantitative comparison of drusen segmented on SD-OCT versus drusen delineated on color fundus photographs. Invest Ophthalmol Vis Sci. 2010 Oct;51(10):4875-83. doi: 10.1167/iovs.09-4962. Epub 2010 Apr 14. PMID 20393117
- [Background] Stopa M, Bower BA, Davies E, Izatt JA, Toth CA. Correlation of pathologic features in spectral domain optical coherence tomography with conventional retinal studies. Retina. 2008 Feb;28(2):298-308. doi: 10.1097/IAE.0b013e3181567798. PMID 18301035
- [Background] Ahlers C, Gotzinger E, Pircher M, Golbaz I, Prager F, Schutze C, Baumann B, Hitzenberger CK, Schmidt-Erfurth U. Imaging of the retinal pigment epithelium in age-related macular degeneration using polarization-sensitive optical coherence tomography. Invest Ophthalmol Vis Sci. 2010 Apr;51(4):2149-57. doi: 10.1167/iovs.09-3817. Epub 2009 Sep 24. PMID 19797228
- [Background] Friberg TR, Huang L, Palaiou M, Bremer R. Computerized detection and measurement of drusen in age-related macular degeneration. Ophthalmic Surg Lasers Imaging. 2007 Mar-Apr;38(2):126-34. doi: 10.3928/15428877-20070301-07. PMID 17396693
- [Background] Munch IC, Ek J, Kessel L, Sander B, Almind GJ, Brondum-Nielsen K, Linneberg A, Larsen M. Small, hard macular drusen and peripheral drusen: associations with AMD genotypes in the Inter99 Eye Study. Invest Ophthalmol Vis Sci. 2010 May;51(5):2317-21. doi: 10.1167/iovs.09-4482. Epub 2009 Dec 10. PMID 20007824
- [Background] Wojtkowski M, Sikorski BL, Gorczynska I, Gora M, Szkulmowski M, Bukowska D, Kaluzny J, Fujimoto JG, Kowalczyk A. Comparison of reflectivity maps and outer retinal topography in retinal disease by 3-D Fourier domain optical coherence tomography. Opt Express. 2009 Mar 2;17(5):4189-207. doi: 10.1364/oe.17.004189. PMID 19259255